CLINICAL TRIAL: NCT00689091
Title: A Prospective, Randomized, Controlled Trial Comparing Bispectral Index Monitoring to Electronic Alerts for Prevention of Awareness During Anesthesia in the General Population
Brief Title: Bispectral Index (BIS) Versus Electronic Alerts in the Prevention of Anesthesia Awareness: the Michigan Awareness Control Study
Acronym: MACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Foundation for Anesthesia Education and Research (Other); American Society of Anesthesiologists (Other); Washington University School of Medicine (Other); University of Chicago (Other); University of Manitoba (Other)
Responsible Party: Principal Investigator, George Mashour, Assistant Professor of Anesthesiology and Neurosurgery, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HUM00013626
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Results first posted 2014-11-17 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2017-11

CONDITIONS: Awareness During General Anesthesia
Keywords: Awareness; BIS Monitor; electronic alerts; minimum; alveolar; concentration
MeSH Terms: interventions — Consciousness Monitors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BIS group (Experimental): This group will have BIS values visible and will receive alerts when the value is >60.
  Interventions: Device: Bispectral Index Monitor
- MAC Alert (Active Comparator): This group will receive an alert if total MAC (including intravenous infusions) is <0.5 age-adjusted.
  Interventions: Device: Electronic MAC alert

INTERVENTIONS:
Device: Bispectral Index Monitor — Comparison of two different alerting protocols. One using the bispectral index monitor and one using the MAC alerting protocols.
  Arms: BIS group
Device: Electronic MAC alert — Comparison of two different alerting protocols. One using the bispectral index monitor and one using the MAC alerting protocols.
  Arms: MAC Alert

SUMMARY:
Awareness during anesthesia is a problem receiving increased attention by patients, clinicians, and the general public. The incidence of intraoperative awareness has been reported to be between 1-2/1000 cases, but recent data suggest that this may be an overestimate. The Bispectral Index (BIS) Monitor is an electroencephalographic method of assessing depth of anesthesia that has been shown in one study to reduce the incidence of awareness during anesthesia in the high-risk population (Myles et al, 2004). In the study of Myles et al, the number needed to treat (NNT) in order to prevent one case of awareness in the high-risk population was 138, with an associated cost of approximately US$2200. Since the NNT and the associated cost of treatment would be much higher in the general population, the efficacy of the BIS monitor in preventing awareness in all anesthetized patients needs to be clearly established. Furthermore, recent data suggest that the BIS may not be useful in the high-risk population. The investigators propose a prospective, randomized, controlled trial comparing the BIS monitor to electronic alerts based on non-electroencephalographic gauges of anesthetic depth.

DETAILED DESCRIPTION:
Electronic alerts have been developed and employed at our institution and have been shown to increase compliance with both clinical and administrative tasks (O'Reilly et al, 2006; Kheterpal et al, 2007). The investigators have developed electronic alerts for the purpose of informing the clinician of potentially insufficient anesthesia based on minimum alveolar concentration (MAC). The algorithm is as follows:

* Every 5 minutes the alerting system checks every active case in our operating rooms. It takes approximately 1 second for this scan of all active cases to occur.
* Conditions for an "active case" are:

  1. data capture is possible (i.e., not a paper record)
  2. data capture is active (i.e., "patient in room" has been electronically entered and end-tidal [Et] CO2 is detected)
  3. case has been identified as a general anesthetic
  4. "anesthesia induction end" has already been documented
  5. request for recovery room bed or transport to an intensive care unit has not been documented
  6. surgical dressing completion has not been documented
* The alerting system checks the most recent value (within a specified time period) of:

  1. Et Sevoflurane (MAC=2.0)
  2. Et Isoflurane (MAC=1.2)
  3. Et Desflurane (MAC=6)
  4. Et Nitrous Oxide (MAC=105) and compares it to the MAC of each agent. It adds the resulting MAC values together for "current total MAC."
* The system then checks for a charted propofol infusion in mcg/kg/min and divides by 150, assuming that 150 mcg/kg/min is "1.0 MAC" for propofol. The analogous concept of MAC for propofol is "Cp50"- the plasma or blood concentrations at which 50% of patients do not move in response to a noxious stimulus. Since the investigators do not have the technology at our institution to calculate Cp50 or Cp50-awake, the investigators have chosen the above propofol dose as an initial value based on clinical experience. The resultant MAC equivalent is added to current total MAC.
* The system next checks for a dexmedetomidine infusion with a rate of 0.2 mcg/kg/hour or greater. If present, it multiplies the current total inhalational MAC by 2, as dexmedetomidine can reduce MAC by 50%.
* At this point, the "current total MAC" is defined as: Et Sevo /2 + Et Iso /1.2 + Et Des/6 + Et Nitrous /105 + propofol rate (in mcg/kg/min)/150. If dexmedetomidine is >0.2 mcg/kg/hour, inhalational MAC is multiplied by 2.
* If this total mac < 0.50, it checks to see if a bolus of propofol, midazolam, etomidate, or thiopental has been given in the preceding 10 minutes.
* It alerts the clinician signed into the case within 30-60 seconds if total age-adjusted MAC < 0.50 AND no bolus has been documented in the last 10 minutes.

This will be the protocol in the MAC-guided group. In the BIS-guided group an electronic alert will be sent if the BIS value is >60. If an alert is triggered, the clinician electronically signed into the case receives an alphanumeric page stating "Potentially insufficient anesthesia, please check vaporizers and intravenous lines."

The investigators are collaborating with Washington University, the University of Chicago, and the University of Mannitoba, who will also be testing a MAC-based protocol in comparison to the BIS.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age, English-speaking, available for follow-up interview at one month.

Exclusion Criteria:

* Pre-existing neurologic or neuropsychiatric condition, surgical manipulation around forehead, not available for follow-up interview.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22185 (Actual)
Dates: Start 2008-05; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George A. Mashour, M.D., Ph.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Medical School, University Hospital, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Vance JL, Shanks AM, Woodrum DT. Intraoperative bispectral index monitoring and time to extubation after cardiac surgery: secondary analysis of a randomized controlled trial. BMC Anesthesiol. 2014 Sep 18;14:79. doi: 10.1186/1471-2253-14-79. eCollection 2014. PMID 25249789
- [Derived] Shanks AM, Avidan MS, Kheterpal S, Tremper KK, Vandervest JC, Cavanaugh JM, Mashour GA. Alerting thresholds for the prevention of intraoperative awareness with explicit recall: a secondary analysis of the Michigan Awareness Control Study. Eur J Anaesthesiol. 2015 May;32(5):346-53. doi: 10.1097/EJA.0000000000000123. PMID 25010744
- [Derived] Avidan MS, Palanca BJ, Glick D, Jacobsohn E, Villafranca A, O'Connor M, Mashour GA; BAG-RECALL Study Group. Protocol for the BAG-RECALL clinical trial: a prospective, multi-center, randomized, controlled trial to determine whether a bispectral index-guided protocol is superior to an anesthesia gas-guided protocol in reducing intraoperative awareness with explicit recall in high risk surgical patients. BMC Anesthesiol. 2009 Nov 30;9:8. doi: 10.1186/1471-2253-9-8. PMID 19948045
- [Derived] Mashour GA, Tremper KK, Avidan MS. Protocol for the "Michigan Awareness Control Study": A prospective, randomized, controlled trial comparing electronic alerts based on bispectral index monitoring or minimum alveolar concentration for the prevention of intraoperative awareness. BMC Anesthesiol. 2009 Nov 5;9:7. doi: 10.1186/1471-2253-9-7. PMID 19891771

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 22,185 patients were recruited but 584 were excluded after recruitment due to change in anesthetic technique, case cancellation, withdrawal, or death. Therefore, 21,601 patients were randomized.
Groups:
- Bispectral Index Group: This group will have BIS values visible and will receive alerts when the value is >60.
  Bispectral Index Monitor: Comparison of two different alerting protocols. One using the bispectral index monitor and one using the MAC alerting protocols.
- Minimum Anesthesia Contration Alert: This group will receive an alert if total MAC (Minimum Anesthesia Concenration) (including intravenous infusions) is <0.5 age-adjusted.
  Electronic MAC alert: Comparison of two different alerting protocols. One using the bispectral index monitor and one using the MAC alerting protocols.
Period: Overall Study
Arm/Group | Bispectral Index Group | Minimum Anesthesia Contration Alert
Started | 10831 | 10770
Completed | 9460 | 9376
Not Completed | 1371 | 1394

BASELINE CHARACTERISTICS:
Groups:
- Minimum Anesthesia Concentration Alert: This group will receive an alert if total MAC (including intravenous infusions) is <0.5 age-adjusted.
  Electronic MAC alert: Comparison of two different alerting protocols. One using the bispectral index monitor and one using the MAC alerting protocols.
- Total: Total of all reporting groups
Arm/Group | Bispectral Index Group | Minimum Anesthesia Concentration Alert | Total
Number analyzed (Participants) | 9,460 | 9,376 | 18836
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 53 [41 to 64] | 53 [41 to 64] | 53 [41 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5,223 | 5,175 | 10398
  Male | 4,237 | 4,201 | 8438

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Incidences With Explicit Recall in the BIS Versus MAC Alert Groups.
Description: By modified intention-to-treat analysis
Time Frame: Outcome of awareness is assessed 30-days after the operation
Measure: Number (95% Confidence Interval); unit: Percentage of participants/30days
Arm/Group | BIS Group | MAC Alert
Number analyzed (Participants) | 9,460 | 9,376
Percentage of participants/30days | 0.08 [0.04 to 0.16] | 0.12 [0.07 to 0.21]

2. Secondary Outcome: Number of Participants With Dreams During Anesthesia Compared Between MAC or BIS Monitoring
Description: Binary variables for whether participants recall dreaming or not.
Time Frame: During surgery (45 minutes - 18 hours), measured based on 30 day interviews
Measure: Count of Participants; unit: Participants
Arm/Group | MAC Alert | BIS Group
Number analyzed (Participants) | 9376 | 9460
Participants
  No dreaming | 9174 | 9352
  Dreaming | 202 | 108

3. Secondary Outcome: Percentage of Cases With Electronic Alerts
Time Frame: During surgery: (45 minutes - 18 hours)
Measure: Mean (Standard Deviation); unit: Percentage of cases
Arm/Group | MAC Alert | BIS Group
Number analyzed (Participants) | 9376 | 9460
Percentage of cases | 2.4 (7.5) | 2.3 (6.6)

4. Secondary Outcome: Overall Use of Anesthetics Comparing the BIS to MAC Alerts.
Time Frame: During surgery (45 minutes - 18 hours)
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | MAC Alert | BIS Group
Number analyzed (Participants) | 9376 | 9460
mg | 0.9 [0.8 to 1.1] | 0.9 [0.8 to 1.1]

5. Secondary Outcome: Time Till Discharge Readiness
Description: measured in time within Post Anesthesia Care Unit ( PACU) until the participant is ready for discharge from PACU based on a composite of factors, including pain and neurologic status
Time Frame: During recovery room stay: 30 minutes to 6 hours
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | MAC Alert | BIS Group
Number analyzed (Participants) | 9376 | 9460
minutes | 98 [66 to 140] | 95 [64 to 138]

6. Secondary Outcome: Number of Participants Without Nausea or Vomiting
Time Frame: During recovery room stay: 30 minutes to 6 hours
Population: Nausea and vomiting numbers were dependent on nurse reporting; as not all nurses did, the participants analyzed are fewer than the total number in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | MAC Alert | BIS Group
Number analyzed (Participants) | 7329 | 4707
Participants
  No nausea: number analyzed (Participants) | 6787 | 4403
  No nausea | 6184 | 4042
  No vomiting | 7149 | 4617

7. Secondary Outcome: Comparison of the Prospective and Retrospective Approaches to the Study Awareness Incidence.
Description: There is controversy regarding the appropriate technique for assessing awareness during anesthesia with explicit recall. A total cohort was utilized to compare the incidence of awareness with recall as determined by formal interview vs. the incidence of awareness with recall based on spontaneous reports (in the same cohort).
Time Frame: 30 days after surgery
Measure: Number; unit: participants
Groups:
- Spontaneous Reporting: any time up to 30 days
- Formal Interview Report: at 30 days
Arm/Group | Spontaneous Reporting | Formal Interview Report
Number analyzed (Participants) | 18836 | 18836
participants
  Yes (awareness with recall) | 3 | 19
  No (no awareness with recall) | 18833 | 18817

8. Other Pre Specified Outcome: Relationship Between BIS Values and Hemodynamic Parameters.
Time Frame: Outcome of hemodynamic stability is assessed
Reporting Status: Not Posted

9. Other Pre Specified Outcome: The Relationship Between Cumulative Deep Hypnotic Time, Anesthetic Doses, and Mortality.
Time Frame: Outcome of mortality is assessed
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Predictors of Post-traumatic Stress Disorder Based on the Type of Awareness Event.
Time Frame: Outcome of post-traumatic stress disorder is assessed with the covariate of awareness
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Anesthetic Induction Doses, Hypotension, and BIS Values.
Time Frame: Outcome of hypotension in relationship to induction doses and BIS values will be assessed
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Meta-Analysis of Awareness Events in Conjunction With the BAG-RECALL Study Based at Washington University.
Time Frame: Outcome of awareness is assessed
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Incidence of Post-traumatic Stress Disorder.
Time Frame: NEED VALUE HERE
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- Miniumum Anesthesia Concentration Alert: This group will receive an alert if total MAC (including intravenous infusions) is <0.5 age-adjusted.
  Electronic MAC alert: Comparison of two different alerting protocols. One using the bispectral index monitor and one using the MAC alerting protocols.
Arm/Group | Bispectral Index Group | Miniumum Anesthesia Concentration Alert
Serious Adverse Events (participants affected / at risk) | 0/9460 | 0/9376
Other Adverse Events (participants affected / at risk) | 0/9460 | 0/9376
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bispectral Index Group (N=9460) | Miniumum Anesthesia Concentration Alert (N=9376)
Non life threatening adverse events (Cardiac disorders) | 0 | 0 — No adverse events resulted from this study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No